CLINICAL TRIAL: NCT06100796
Title: Effect of Diabetes Mellitus on Outcomes and Response Rate in Patients With Advanced NSCLC on Immunotherapy
Brief Title: Effect of DM on Outcomes and Response Rate in Patients With Advanced NSCLC on ICI
Acronym: NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Momen Gebril Reyad Eltaher, Assistant lecturer, Assiut University
Other Study IDs: ICI outcomes in NSCLC with DM
Record Dates: First submitted 2023-10-14; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Diabetes Mellitus
Keywords: NSCLC; DM; ICI; OHA
MeSH Terms: conditions — Diabetes Mellitus | interventions — pembrolizumab; Hypoglycemic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Pembrolizumab — Immune check inhibitor with OHA
  Other Names: oral hypoglycemic agents

SUMMARY:
Retrospectively investigating the effect of DM on response rate and outcomes during immunotherapy treatment in patients with NSCLC in the last 5 years.

DETAILED DESCRIPTION:
Lung cancer continues to be the most common cause of cancer-related death worldwide for both males and females despite the identification of clinically-actionable driver mutations in genomic subgroups of patients. Non-small cell lung cancer (NSCLC) is the most common histological diagnosis for 85% of lung cancer patients. Immune checkpoint inhibitors (ICI) has significantly altered the prognosis for patients with advanced non-small cell lung cancer (mNSCLC) as it has been shown to have distinct and long-lasting impacts on survival in first and second line treatment. As a result, immunotherapy has emerged as the backbone of care for people with NSCLC. Although some patients benefit considerably from ICI, not all patients do. A comprehensive research effort exists to identify and characterize variables that could predict or boost the response to ICI.

At the same time, diabetes mellitus (DM) is becoming more prevalent globally and lung cancer patients frequently suffer from a variety of comorbidities, including (DM). However, its effect on treatment outcomes is still unclear, particularly in the era of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with advanced Non Small Cell Lung Cancer who received Immune Check Inhibitors alone or in combination with chemotherapy, either as first line or as a subsequent line

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All available patients from 2018 till December 2023 will be included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 12 weeks after starting immunotherapy regimen.
  CT evaluation for response rate measured by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Ali Gamal, Study Chair — Assistant Lecturer
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided